CLINICAL TRIAL: NCT06812520
Title: Educational Intervention to Promote Compression Therapy in People With Venous Ulcer: Pilot and Non-randomized Feasibility Study
Brief Title: Educational Intervention to Promote Compression Therapy in People With Venous Ulcer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alide Salazar Molina (Other)
Responsible Party: Sponsor-Investigator, Alide Salazar Molina, Ingrid Briones Luengo, Universidad de Concepcion
Organization: Universidad de Concepcion (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CEBB1659-2024
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Varicose Ulcer
Keywords: Varicose ulcer; adherence; Patient education; Acceptability
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: A feasibility study will be carried out. For this purpose, a study will be carried out without a control group with a pre- and post-test comparison, since it corresponds to phase I of development of an intervention study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Educational intervention group for adherence (Experimental): The study only has the intervention group who will receive the educational activity to improve adherence to compression therapy.
  Interventions: Behavioral: Educational intervention in adherence

INTERVENTIONS:
Behavioral: Educational intervention in adherence — An educational intervention of 4 face-to-face sessions will be carried out as a complement to the care provided by professionals to users with venous ulcers, which consists of the advanced healing procedure that includes compressive bandaging of the venous ulcer.

SUMMARY:
Background: Chronic Venous Disease (CVD) is a condition that affects a significant percentage of the world's population, and can range from mild symptoms such as telangiectasias to severe manifestations such as venous ulcers (VU). The gold standard UV treatment is compression therapy, however, people's adherence to it is variable due to several associated factors: physical, aesthetic and lack of education about compression therapy. Compression therapy acts by increasing interstitial pressure, thus decreasing the caliber of superficial and deep veins, decreasing venous pressure and edema . The study originates from clinical practice where it is observed that people do not adhere or abandon compression treatment, a situation that agrees with the literature review, so new trials on strategies to increase adherence are required (20). The proposed intervention: promoting adherence has a theoretical basis, a conceptual basis and an empirical basis. a) Theoretical basis: it incorporates the theory of self-care of chronic diseases with the incorporation of symptoms, due to the importance that these have for those who present them and for the self-care process, particularly with regard to maintaining self-care and adherence; in addition, the theoretical basis related to health interventions is incorporated. b) Conceptual basis: founded on vascular alterations that lead to the loss of skin integrity with the consequent imbalance: pain, edema, exudate, bad odor, so it is necessary for these to be recognized by patients and then by the professionals who serve them. c) Empirical basis: it incorporates compression therapy, considered the gold standard in the treatment of people with venous ulcers. Based on the evidence analyzed, the Lively Leg intervention developed by Heinen et al. was chosen as a basis. 2012, to which modifications were introduced based on the self-care theory, since, together, the symptoms of the ulcer, the associated chronic diseases and the characteristics of the people intervene in their adherence to compression therapy. The objective of the study is to evaluate the feasibility and preliminary effect of an educational intervention on adherence to compression therapy, pain and ulceration of the area in users who have a venous ulcer, in the commune of Hualpen, Chile, during the year 2024.

DETAILED DESCRIPTION:
Type of study design A feasibility study will be carried out. For this purpose, a study will be carried out without a control group with a pre- and post-test comparison, since it corresponds to phase I of development of an intervention study.

Study hypotheses.

* Users who have a venous ulcer and compression therapy, after the educational intervention, have a smaller area of ulceration than at the beginning of the intervention.
* 50% of users who present venous ulcer and compression therapy show adherence to therapy after the educational intervention.
* Users who have a venous ulcer and compression therapy, after the educational intervention, have a lower intensity of pain than at the beginning of the intervention.
* Users who present with venous ulcer and compression therapy evaluate the acceptability of an educational intervention with a score greater than 2.

who can participate? People over 20 years of age who have a venous ulcer, registered in the commune of Hualpen who meet the inclusion and exclusion criterio.

What are possible risks and benefits of participating? The main risk is presenting some psychoemotional alteration due to possible experiences and experiences or simply not wanting to continue, which would constitute a sufficient reason to suspend the interview, and if psychoemotional symptoms are presented, crisis care will be provided and then referred to the health Center, for your attention and which would constitute sufficient reason to suspend the interview.

The benefits of participation involve all those that are associated with ulcer healing: decrease or closure of the ulcer, decrease in pain, decrease in wound exudate, increase in control of symptoms and signs of venous ulcer, less quantity of cures, improve quality of life, greater mobility.

Patient recruitment will be carried out for convenience; the number of participants to be entered is 22, which was calculated with an estimated loss of 20%.

Recruitment of users will begin in December and is estimated to take place over 2 to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a grade 2 venous ulcer who is admitted to compression treatment
* Alphabet.
* Management of the Spanish language

Exclusion Criteria:

* Adult who presents a grade 1 venous ulcer
* Adult who presents cognitive impairment (determined by review of clinical record by treating nurse)
* Diagnoses of: dementia,
* Diagnoses Alzheimer's disease
* mental retardation or cognitive deficit
* Adult with severe dependency (determined by review of clinical record by treating nurse) Adult with venous ulcer with cancer undergoing chemotherapy (determined by review of clinical record by treating nurse.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability assessment will be carried out by applying the TAP scale | 12 weeks
  Acceptability will be measured through the Questionnaire developed by Sidani "Treatment Acceptability and Preference" (TAP) adapted to Chilean Spanish.
  A total scale score is computed as the mean of the four items' scores to reflect level of perceived treatment acceptability. The possible range for the total scale score is 0 to 4, with high score reflecting high acceptability
Adherence to compression therapy | 12 weeks
  Adherence can be defined as the degree to which patients follow the instructions given to them by different professionals. In this study, adherence to compression therapy will be assessed on each occasion that they attend visits and those who have a percentage of adherence to therapy equal to or above 75% in the 12-week period will be categorized as adherent.
area of ulceration | 12 weeks
  Surface of the wound that is open, the evaluation is carried out by measuring in centimeters the length at its greatest and width at its largest ends and then multiplying both, with this the ulceration area is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Alide A Salazar, Doctor, Study Director — Universidad de Concepcion
Locations (1):
- Departamento de Salud de la comuna de Hualpen, Hualpén, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: No